CLINICAL TRIAL: NCT03636035
Title: Assessment of Performance of Participants With Mild Knee Osteoarthritis Taking Tregocel® as a Dietary Supplement Alongside Standard of Care Treatment
Brief Title: Tregocel® as a Dietary Supplement in Mild Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Biocare Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MBTR01
Record Dates: First submitted 2018-08-08; First posted 2018-08-17 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2020-02

CONDITIONS: Mild Knee Osteoarthritis
Keywords: dietary supplement; arthritis; joint; complementary medicine
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tregocel® supplementation (Experimental): Tregocel® coated tablets (2/day) orally for 36 weeks
  Interventions: Dietary Supplement: Tregocel®

INTERVENTIONS:
Dietary Supplement: Tregocel® — Coated tablet (oral)

SUMMARY:
This study is an assessment of the overall performance of participants with symptomatic mild knee OA taking Tregocel® as a dietary supplement in addition to standard of care treatment.

DETAILED DESCRIPTION:
Tregocel® is a combination herbal product which as a dietary supplementation may help maintain proper performance of joints. Although some studies have reported beneficial effects for individual components of Tregocel®, there have been no clinical assessments of supplementation with Tregocel® as a finished product. This study will involve collection of data on Tregocel® supplementation in participants with symptomatic mild knee osteoarthritis (OA) who are already receiving standard pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with all study procedures
* Fulfilment of consent process
* Documented diagnosis of radiologically confirmed mild knee osteoarthritis with stable pain management (including patello-femoral joint, Kellgren-Lawrence classification ≤2 and clinical symptoms lasting more than 6 months prior to screening)
* Maximal pain score ≥30 on a 100 mm VAS at screening and confirmed at baseline, with PRN use of analgesics during run-in
* Completed patient diary during run-in
* Ambulant with ECOG score <2

Exclusion Criteria:

* pregnancy or breastfeeding (women)
* body mass index less than 18.5 kg/m^2 or more than 35.0 kg/m^2.
* secondary knee OA
* clinically apparent tense effusion of the target knee
* valgus/varus knee/foot deformities, ligament laxity, or meniscal instability
* changes in regular OA therapy during screening
* chronic diseases which may require treatment with systemic steroids
* progressive serious medical conditions
* severe organ dysfunction
* cardiac insufficiency
* history of gastrointestinal ulcer or bleeding.
* any significant medical conditions that may interfere with the study procedures, safety, compliance or overall participation in the study
* allergies or intolerance to any of the dietary supplement ingredients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in distance walked in 6-minutes as an indicator of AMBULATORY MOBILITY | Tested at Baseline (week 0) and at end of supplementation (week 36)
  Challenge involves subject walking unimpeded along a continuous straight line of 30 metre in distance with no incline. Distance covered will by an assistant sured with a 30 metre metric tape measure. Laps and time will be tracked manually with a digital lap counter and timer (second). Baseline values will be compared to values after supplementation to determine any change in individual performance.

SECONDARY OUTCOMES:
Physical exam parameter 1: BODY WEIGHT measurement | Screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Body weight measure using digital scales (recorded in kilogram).
Physical exam parameter 2: SUBJECT HEIGHT measurement | Screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Body height measured manually using a wall tape measure (recorded in metre). Weight and height values will be used to calculate body mass index [weight (kilogram) / height (metre) ^2]
Vital sign 1: BODY TEMPERATURE | Screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Measured using a digital ear thermometer after 5 minutes rest, sedentary.(recorded in degree Celsius)
Vital sign 2: BLOOD PRESSURE | Screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Systolic and diastolic blood pressure values will be determined using an automated sphygnomanometer after 5 minutes rest, sedentary (recorded in millimeter mercury).
Vital sign 3: PULSE RATE | Screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Recorded using an automated sphygnomanometer after 5 minutes rest, sedentary (beats / minute)
Arthritis self-assessment 1: Initial degree of PERCEIVED PAIN represented by manual marking on a simplified printed 100mm linear scale (during Run-in) | Run-in period (week -1 to week 0)
  Subject responds to a request to report maximal pain experienced in 48 hours in target knee by pen or pencil marking along a 100mm line scale (0mm (left) = no pain; 100mm (right) = extreme pain; marks closer to right indicate more pain). Length from 0mm to mark will be measured using a 300mm ruler, to indicate the degree of maximal pain felt. No subscales are included in this assessment. Marks appearing between centre of the line and 100mm limit are considered moderate to severe (total score range = 0-100mm)
Arthritis self-assessment 2: change in degree of PERCEIVED PAIN represented by manual marking on a printed 100mm linear scale (During and after supplementation) in response to WOMAC questionnaire | Scores taken at baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Subject responds to a request to report degree of pain experienced in 48 hours in target knee by pen or pencil marking along a 100mm horizontal line (0mm (left) = no pain; 100mm (right) = extreme pain; more pain = closer to right hand end of line). Length from 0mm to mark will be measured using a 300mm ruler. Report includes degree of pain felt while stationary or during normal movement (a set of 5 subscales appearing as separate lines with the same limits). Marks appearing between the centre of the line and 100mm limit are considered between moderate and severe, with more severe toward the right. Total score is a sum of the 5 subscales (range 0-500mm). WOMAC = Western Ontario and McMaster Universities Arthritis index.
Arthritis self-assessment 3: change in degree of PERCEIVED STIFFNESS represented by manual marking on a printed 100mm linear scale (During and after supplementation) in response to WOMAC questionnaire. | Scores taken at baseline (0 week); rescored at 12, 24, 36 and 40 weeks
  Subject responds to a request to report feeling of stiffness experienced in 48 hours in target knee by pen or pencil marking along a 100mm horizontal line (0mm (left) = no stiffness; 100mm (right) = extreme stiffness; more pain = closer to right hand end of line). Length from 0mm to mark will be measured using a 300mm ruler, to indicate the degree of stiffness felt at start and end of a day (a set of 2 subscales, appearing as separate lines with the same limits). Marks appearing from the centre of the line to 100mm limit are considered between moderate and severe, with more severe toward the right. Total score is a sum of the 2 subscales (range 0-200mm).
Arthritis self-assessment 4: change in degree of PERCEIVED DIFFICULTY WITH DAILY TASKS represented by manual marking on a printed 100mm linear scale (During and after supplementation) in response to WOMAC questionnaire. | Scores taken at baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Subject responds to a request to report difficult in performing daily tasks in 48 hours due to arthritis in target knee by pen or pencil marking along a 100mm horizontal line (0mm (left) = no pain; 100mm (right) = extreme pain; more pain = closer to right hand end of line). Length from 0mm to mark will be measured using a 300mm ruler, to indicate the degree of difficulty experienced in different domestic activities (set of 17 subscales, appearing as separate lines with the same limits). Marks appearing between the centre of the line to 100mm limit are considered between moderate and severe, with more severe toward the right. Total score is a sum of the 17 subscales (range 0-1700mm).
Change in target KNEE FLEXIBILITY assessment, based on heel-thigh distance and knee angle at maximal flexion. | Scores taken supine and prone for both knees at baseline (week 0); rescored at 12, 24, 36 weeks
  Subjects will lie either supine or prone while holding their target knee statically as close to their thigh as is bearable. Distance from heal to thigh (standard tape measurement) and angle of knee (measured using a goniometer) will be recorded.
Safety assessment 1: clinical HEMATOLOGY parameters (a) Blood cell count | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Number erythrocytes leukocytes and platelets initially and changes thereafter determined using an automated blood sample analyser (number x 10^9/litre)
Safety assessment 1: clinical HEMATOLOGY parameters (b) hemoglobin level | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Hemoglobin will be measured initially and any subsequent changes determined using UV/Vis spectrometry (g/dL).
Safety assessment 1: clinical HEMATOLOGY parameters (c) sodium level | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Blood sodium initially and any subsequent changes to be determined using a blood gas analyser (mM)
Safety assessment 1: clinical HEMATOLOGY parameters (d) potassium level | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Blood sodium initially and any subsequent changes to be determined using a blood gas analyser (mM)
Safety assessment 1: clinical HEMATOLOGY parameters (e) aspartate alanine transferase level | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Blood aspartate alanine transferase initially and any subsequent changes to be determined using ELISA assay (IU/L)
Safety assessment 1: clinical HEMATOLOGY parameters (f) alanine aminotransferase | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Blood alanine aminotransferase level initially and any subsequent changes to be determined using ELISA assay (IU/L)
Safety assessment 1: clinical HEMATOLOGY parameters (g) total bilirubin level | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Blood bilirubin initially and any subsequent changes to be determined using ELISA assay (IU/L).
Safety assessment 1: clinical HEMATOLOGY parameters (h) alkaline phosphatase level | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Alkaline phosphatase level initially and any subsequent changes to be determined using ELISA assay (IU/L).
Safety assessment 1: clinical HEMATOLOGY parameters (i) creatine level | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Creatine level initially and any subsequent changes to be determined using ELISA assay (IU/L).
Safety assessment 1: clinical HEMATOLOGY parameters (j) blood sodium | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Sodium level initially and any subsequent changes to be determined using a blood gas analyser (mM).
Safety assessment 1: clinical HEMATOLOGY parameters (k) blood potassium | Performed at screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Potassium level initially and any subsequent changes to be determined using a blood gas analyser (mM).
Safety assessment 2: URINALYSIS (a) presence of leukocytes | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (negative = grey, positive = increase in purple color intensity).
Safety assessment 2: URINALYSIS (b) presence of nitrites | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (negative = yellow, positive = increase in pink color intensity).
Safety assessment 2: URINALYSIS (c) level of urobilinogen | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (normal = 0.2-1 mg/dL, yellow; raised = 2-8 mg/dL, with increasing pink intensity).
Safety assessment 2: URINALYSIS (d) presence of protein | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (none or trace amounts (quince); raised = increased darkness of green pigment)
Safety assessment 2: URINALYSIS (e) pH | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (dual pigment assay, represented by color change from fading of orange (pH 5) to increased darkness of green pigment (pH 8.5).
Safety assessment 2: URINALYSIS (f) presence of blood | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (none = yellow; trace amounts of non-hemolysed blood (dark-green speckle discoloration on a yellow background); presence of hemolysed blood (increasing darkness of green pigment on yellow background).
Safety assessment 2: URINALYSIS (g) specific gravity (SG) | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (Dark green = 1.000, yellow-green = 1.030; increasing SG correlates with decreasing darkness of green pigment.
Safety assessment 2: URINALYSIS (h) ketone level | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (none = beige; trace (pink = 5, increasing to large (160) mg/dL with increasing darkness of burgundy pigment)
Safety assessment 2: URINALYSIS (i) presence of bilirubin | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested initially and any subsequent changes determined colorimetrically (negative = yellow; increasing levels correlate with appearance of light brown pigment).
Safety assessment 2: URINALYSIS (j) glucose level | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested and measured, and subsequent changes determined colorimetrically for content of glucose (absence = blue-green; presence = range form 100 (green) to > 2000 mg/dL (dark brown).
Safety assessment 2: URINALYSIS (k) presence of human chorionic gonadotrophin (hCG) | Performed at screening (week -2), baseline (Week 0); rescored at 12, 24, 36 and 40 weeks
  Urine will be dipstick tested and measured colorimetrically for presence of hCG (positive test = appearance of blue line on white background; negative = remains white).
Determination of total usage of PRESCRIPTION ANALGESICS | Screening (week -2), baseline (week 0); rescored at 12, 24, 36 and 40 weeks
  Usage of any analgesics will be recorded on a daily basis by subjects using diary, which will be reviewed at clinical consultation. Total consumption will be logged at the end of the supplemention period as an indicator of changes in reliance on prescribed medications. (expressed as number of medications per day, regardless of type).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Wilczek, MD, Principal Investigator — Coramed, Wroklaw
Locations (1):
- Clinmed Pharma, Warsaw, Poland

REFERENCES:
- [Derived] Zegota Z, Gozdzik J, Glogowska-Szelag J. IMPROVED PHYSICAL FUNCTION WITH COMPLEMENTARY USE OF A DIETARY SUPPLEMENT FOR MILD KNEE OSTEOARTHRITIS: A SUBGROUP ANALYSIS. Wiad Lek. 2021;74(9 cz 1):2128-2137. PMID 34725289